CLINICAL TRIAL: NCT02226783
Title: Phase I Study in Healthy Subjects to Evaluate the Pharmacodynamics (PD) of AZD1722 Given With and Without Food (Part A) and a 2-way Crossover to Evaluate the PD of AZD1722 Given as a Free-base Tablet With and Without Omeprazole (Part B)
Brief Title: D5611C00003 - Food Interaction Study With AZD1722 Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5611C00003
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers Food Interaction Study
Keywords: Phase I; Healthy subjects; PK; PD
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment A AZD1722 salt tablet (fasted) (Experimental): Part A-Treatment A: morning dose of AZD1722 salt tablet 5 to 10 minutes before start of intake of breakfast; evening dose 5 to 10 minutes before start of intake of dinner
  Interventions: Drug: AZD1722 salt tablet
- Treatment B AZD1722 salt tablet (fed) (Experimental): Part A Treatment B: morning dose of AZD1722 salt tablet 30 minutes after start of intake of breakfast; evening dose 30 minutes after start of intake of dinner
  Interventions: Drug: AZD1722 salt tablet
- Treatment C AZD1722 salt tablet (fasted) (Experimental): Part A Treatment C: morning dose AZD1722 HCl tablet then breakfast served 1 hour after dosing; evening dose 3 hours after start of intake of dinner and 1 hour before the next meal consumption
  Interventions: Drug: AZD1722 salt tablet
- Treat D AZD1722 free-base tablet (fast) (Experimental): Part B Treatment D: morning dose of AZD1722 free-base tablet administered 5 to 10 minutes before the start of intake of breakfast and evening dose 5 to 10 minutes before start of intake of dinner
  Interventions: Drug: AZD1722 free base tablet
- Treat E AZD1722 free-base+Omeprazole (Experimental): Part B Treatment E: morning dose of AZD1722 free base tablet administered 5 to 10 minutes before start of intake of breakfast and evening dose 5 to 10 minutes before start of intake of dinner; omeprazole was administered twice daily from Days -5 to -1 or Days 5 to 9 (depending on assigned treatment period), 1 hour before breakfast and dinner, and from Days 1 to 4 or Days 10 to 13, 1 hour prior to the administration of AZD1722
  Interventions: Drug: AZD1722 free base tablet; Drug: AZD1722 free base tablet + Omeprazole

INTERVENTIONS:
Drug: AZD1722 salt tablet — AZD1722 will be administered as 14 mg (salt tablet). tablet for oral use. Subjects will receive a 14 mg tablet in the morning and evening on Days 1 to 4 (Period 1), Days 7 to 10 (Period 2), and Days 13 to 16 (Period 3).
  Arms: Treatment A AZD1722 salt tablet (fasted); Treatment B AZD1722 salt tablet (fed); Treatment C AZD1722 salt tablet (fasted)
Drug: AZD1722 free base tablet — AZD1722 will be given as four 14 mg free-base tablets (56mg) in the morning and evening on Days 1 to 4 (Period 1) and Days 10 to 13 (Period 2).
  Arms: Treat D AZD1722 free-base tablet (fast); Treat E AZD1722 free-base+Omeprazole
Drug: AZD1722 free base tablet + Omeprazole — AZD1722 free base tablet administered 5 to 10 minutes before intake of breakfast and evening dose 5 to 10 minutes before start of intake of dinner; omeprazole was administered twice daily from Days -5 to -1 or Days 5 to 9 (depending on assigned treatment period), 1 hour before breakfast and dinner, and from Days 1 to 4 or Days 10 to 13, 1 hour prior to the administration of AZD1722
  Arms: Treat E AZD1722 free-base+Omeprazole

SUMMARY:
Study to evaluate the effect of intake of food in comparison to fasting condition on pharmacodynamics of AZD1722 following a twice-daily administration of AZD1722 tablet formulation

DETAILED DESCRIPTION:
A Phase I, Open-label, Randomized, Single-center, 3-way Crossover Study in Healthy Subjects to Evaluate the Pharmacodynamics Effects of AZD1722 Administered With and Without Food (Part A) plus a 2-way Crossover in Subjects to Evaluate the Pharmacodynamic Effect of AZD1722 Administered as an AZD1722 Free-base Tablet with and without Omeprazole (Part B)

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers aged 18 to 65 years
2. Females of childbearing potential had to have a negative pregnancy test and females of childbearing potential included in the study had to use 2 effective methods of avoiding pregnancy, females of nonchildbearing potential to fulfill 1 of the following criteria:

   1. Postmenopausal, defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatment and luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range
   2. Documentation of irreversible surgical sterilization by hysterectomy, tubal occlusion, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation
3. Had a body mass index (BMI) of 18 and 30 kg/m2, inclusive, and weight at least 50 kg and no more than 100 kg
4. Regular bowel habits of at least 1 stool portion per day.

Exclusion Criteria:

(1) History of clinically-significant disease or disorder (2) History or presence of GI, hepatic, or renal disease, including GI surgery, or any condition known to interfere with absorption, distribution, metabolism, or excretion of drugs. (3) Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks (4) any clinically-significant abnormalities in clinical chemistry, hematology, or urinalysis.

(5) Abnormal vital signs after a 10-minute supine rest, any clinically-significant abnormalities in rhythm, conduction, or morphology of resting ECG (6) Prolonged QTcF greater than 450 ms or shortened QTcF less than 340 ms or family history of long QT syndrome.

(7) Loose stools (Bristol Stool Form Score [BSFS] of 6 or 7) 2 or more days during the 7 days prior to randomization (8) Use of medications that are known to affect stool consistency and/or GI motility, including fiber supplements, probiotic supplements, probiotic supplements in medication form, antidiarrheals, prokinetic drugs, enemas, probiotic medications or supplements (ie, Activia®); or salt or electrolyte supplements containing sodium, potassium, chloride, or bicarbonate formulations during the past 7 days before randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic:- To evaluate the effect of intake of food in comparison to fasting condition on PD of AZD1722 following a twice-daily administration of AZD1722 tablet formulation | Stool samples will be collected over 24 hr periods from day -2 to Day 17
  Sodium and phosphorus content in stool collected over 24-hour intervals

SECONDARY OUTCOMES:
Pharmacodynamic:- To evaluate the effect of intake of food in comparison to fasting condition on PD of AZD1722 following twice-daily administration of an AZD1722 tablet formulation | Stool samples will be collected over 24 hr periods from day -2 to Day 17
  Stool consistency, weight, and frequency measured on a daily basis
Pharmacodynamic:- To evaluate the effect of intake of food in comparison to fasting condition on PD ofAZD1722 following twice-daily administration of an AZD1722 tablet formulation | Urine will be collected in 24 hour intervals from Day -2 to Day 17
  Urinary sodium and phosphorus content over 24-hour intervals
Pharmacokinetic: To evaluate the plasma concentrations of AZD1722 | Predose, 1, 2, and 4 hours post morning dose for measurement of AZD1722 in plasma will be taken on days 1, 4, 7, 10, 13, and 16
  AZD1722 plasma concentrations

OTHER OUTCOMES:
Safety:- To evaluate the safety of AZD1722 | Safety assessments will be performed throughout the study from Baseline to final follow-up visit (Day-2 to Day 26)
  Adverse events, vital signs, physical examinations, ECGs, and laboratory assessments (chemistry, hematology, and urinalysis)
Exploratory:-To evaluate the effect of high and low gastric pH on the PD of AZD1722 following twice daily administration of an AZD1722 free-base tablet formulation given with and without omeprazole | Stool and urine samples will be collected over 24 hr periods from day -2 to Day 14
  Stool sodium and phosphorus content; stool frequency, weight, and consistency; and urine sodium and phosphorus content assessed over 24-hour intervals

CONTACTS AND LOCATIONS:
Overall Officials: David Mathews, MD, Principal Investigator — Quintiles Phase I Services, LLC
Locations (1):
- Research Site, Overland Park, Kansas, United States